CLINICAL TRIAL: NCT03138616
Title: The Impacts of Vitamin D Supplementation on Glucose Metabolism in Chinese Women With Vitamin D Deficiency and Former Gestational Diabetes Mellitus:A Randomised Control Trial
Brief Title: The Impact of Vitamin D Supplementation on Glucose Metabolism in Chinese Women With Former Gestational Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yufan Wang, Principal Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160901
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational diabetes mellitus; vitamin D; postpartum
MeSH Terms: conditions — Diabetes, Gestational | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: intervention group and control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- vitamin D intervention group(NGR) (Experimental): normal glucose regulation group according to the oral glucose tolerance test (OGTT) around 42 days postpartum.
  took 1600 units of vitamin D daily for nine months and meanwhile receive lifestyle intervention.
  Interventions: Drug: vitamin D
- control group(NGR) (No Intervention): normal glucose regulation group according to the oral glucose tolerance test (OGTT) around 42 days postpartum.
  only receive lifestyle intervention.
- vitamin D intervention group(IGR) (Experimental): impaired glucose regulation group according to the oral glucose tolerance test (OGTT) around 42 days postpartum.
  took 1600 units of vitamin D daily for nine months and meanwhile receive lifestyle intervention.
  Interventions: Drug: vitamin D
- control group(IGR) (No Intervention): impaired glucose regulation group according to the oral glucose tolerance test (OGTT) around 42 days postpartum.
  only receive lifestyle intervention.

INTERVENTIONS:
Drug: vitamin D — take 1600 units of vitamin D daily for nine months
  Arms: vitamin D intervention group(IGR); vitamin D intervention group(NGR)

SUMMARY:
Vitamin D deficiency are related to insulin resistance and impaired beta-cell function.It is reported that the level of vitamin D is lower during pregnancy and postpartum in the women with Gestational Diabetes Mellitus. The investigators hypothesize that vitamin D supplementation to women after birth with previous gestational diabetes may improve glucose metabolism.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is defined as any degree of glucose intolerance that is first identified during pregnancy, excluding diabetic patients diagnosed before pregnancy. GDM can not only have an adverse effect on the pregnant women and the developing fetus, but also can have long lasting effects after birth. GDM can elevates risks of abnormal glucose metabolism postpartum. Vitamin D deficiency has been shown to be associated with insulin resistance and impaired β-cell function. Our previous research also implied that the level of vitamin D is much lower in the women of impaired glucose regulation after birth with history of GDM. This prospective randomized, control clinical trial was designed to evaluate the effects of vitamin D administration on insulin resistance and β-cell function among women with vitamin D deficiency（25OHD <50 ng/mL）and previous GDM. Participants with vitamin D deficiency and previous GDM were divided into normal glucose regulation group(NGR) (n=90) and impaired glucose regulation group(IGR)(n=90) according to the oral glucose tolerance test (OGTT) around 42 days postpartum. And each group was further divided into intervention group and control group, Participants in the intervention group took 1600 units of vitamin D daily for nine months and meanwhile receive lifestyle intervention. The control group only receive lifestyle intervention. This study aimed to evaluate the impact of vitamin D supplementation on insulin sensitivity, pancreatic β-cell function and markers of inflammation in Chinese women with former GDM and vitamin D insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. with previous GDM,40-50 days after birth -
2. with deficiency of vitamin D(25-(OH)D3<50nmol/L)

Exclusion Criteria:

1. type 1 diabetes，type 2 diabetes and other type of diabetes
2. server disfunction of liver and kidney（ALT >100U/L，Cr>132ummol/L）
3. with mental disease,sever anemia,sever infection,sever heart disease,now is taking asprin, immunosuppressive agent,Antiepileptic drugs
4. pregnancy or plan to pregnant in one year
5. can't understand the requirement of this study
6. disfunction of thyroid

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants with vitamin D deficiency and previous GDM
Enrollment: 180 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in glucose metabolism | 9 months
  change in Insulin sensitivity index,insulin resistance,inflammatory factors

SECONDARY OUTCOMES:
change in Lipid metabolism | 9 months
  change in triglyceride,cholesterol,HDL,LDL and FFA（free fatty acid）
change in metabolism of calcium and phosphorus | 9 months
  change in calcium, phosphorus,the ratio of urine calcium and creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First People's Hospital, Shanghai Jiao Tong University 100 Haining Road,Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nsiah-Kumi PA, Erickson JM, Beals JL, Ogle EA, Whiting M, Brushbreaker C, Borgeson CD, Qiu F, Yu F, Larsen JL. Vitamin D insufficiency is associated with diabetes risk in Native American children. Clin Pediatr (Phila). 2012 Feb;51(2):146-53. doi: 10.1177/0009922811417290. Epub 2011 Oct 20. PMID 22019791
- [Background] von Hurst PR, Stonehouse W, Coad J. Vitamin D supplementation reduces insulin resistance in South Asian women living in New Zealand who are insulin resistant and vitamin D deficient - a randomised, placebo-controlled trial. Br J Nutr. 2010 Feb;103(4):549-55. doi: 10.1017/S0007114509992017. Epub 2009 Sep 28. PMID 19781131
- [Background] Mitri J, Dawson-Hughes B, Hu FB, Pittas AG. Effects of vitamin D and calcium supplementation on pancreatic beta cell function, insulin sensitivity, and glycemia in adults at high risk of diabetes: the Calcium and Vitamin D for Diabetes Mellitus (CaDDM) randomized controlled trial. Am J Clin Nutr. 2011 Aug;94(2):486-94. doi: 10.3945/ajcn.111.011684. Epub 2011 Jun 29. PMID 21715514
- [Background] Pleskacova A, Bartakova V, Pacal L, Kuricova K, Belobradkova J, Tomandl J, Kankova K. Vitamin D Status in Women with Gestational Diabetes Mellitus during Pregnancy and Postpartum. Biomed Res Int. 2015;2015:260624. doi: 10.1155/2015/260624. Epub 2015 Apr 27. PMID 26000285